CLINICAL TRIAL: NCT07155733
Title: Comparison Of The Effectiveness Of Myofascial Release Exercises and Vagus Nerve Neuromodulation in Tinnitus Patients: Randomized Controlled Trial
Brief Title: tVNS and Myofascial Release in Tinnitus
Acronym: TVNS-TINN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Maria SARIKIR, Bsc, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23069
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Chronic Tinnitus; Subjective Tinnitus; Neuromodulation
Keywords: tinnitus; chronic tinnitus; subjective tinnitus; vagus nerve stimulation; Transcutaneous Vagus Nerve Stimulation (tVNS); Auricular Vagus Nerve Stimulation; Neuromodulation; Myofascial Release; Physical Therapy
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Intervention Model Description: This is a three-arm, parallel group randomized controlled trial comparing the effects of transcutaneous vagus nerve stimulation (tVNS), myofascial release exercise, and standart medical care on chronic subjective tinnitus. Participants are randomly assigned to one of three groups and receive their assigned intervanetion to evaluate changes in tinnitus severity, sleep quality and audiometric measures.
Masking Description: This is an open-label study. Both participants and treating clinicians are not blinded due to the nature of the interventions. Outcome assesor who scoring THI, recording VAS, PSQI is not blinded, those who scores audiometric outcomes are blinded to group assignment to reduce assesment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transcutaneous Vagus Nerve Stimulation (Experimental): 10 sessions over 3 weeks; auricular stimulation of the vagus nerve using TENS; session duration 30 min.
  Interventions: Device: Transcutaneous Vagus Nerve Stimulation; Other: Standard medical treatment
- Myofascial Exercise Group (Experimental): 10 supervised sessions over 3 weeks; targeting cervical muscles.
  Interventions: Behavioral: Myofascial Release Exercises; Other: Standard medical treatment
- Control Group (No Intervention): Standart Medical Care without additional inerventions

INTERVENTIONS:
Device: Transcutaneous Vagus Nerve Stimulation — Participants receive 10 sessions of transcutaneous vagus nerve stimulation over 3 weeks using a TENS device. stimulation is applied to the auricular branch of the vagus nerve (cymba conchae/tragus) for 30 minutes per session. Participants continue usual medical care. Parameters (frequency, pulse width, intencity) are standartized according to safety guidelines. This intervention specifically targets the auricular branch of the vagus nerve, distinguishing it from other device-based intervention such as conventional TENS for pain management or non-auricular vagus stimulation used in other studies.
  Arms: Transcutaneous Vagus Nerve Stimulation
Behavioral: Myofascial Release Exercises — Participants receive 10 supervised session over 3 weeks focusing on myofascial release of cervical muscles. in addition to their usual medical management for tinnitus. Exercises are designed to reduse muscle tensionpotentially contributing to tinnitus. This intervention is distinct from general physical therapy or standart relaxation exercises beacause it specifically targets myofascial structures implicated in tinnitus pathophysiology.
  Arms: Myofascial Exercise Group
Other: Standard medical treatment — Participants continue their usual medical management for tinnitus without additional interventions. This group serves as a control to compare the effects of tVNS and myofascial exercises. It differs from sham or placebo interventions used in oter studies because no active or stimalated treatment is provided.
  Arms: Myofascial Exercise Group; Transcutaneous Vagus Nerve Stimulation

SUMMARY:
This randomized controlled trial aims to investigate the effectiveness of transcutaneous vagus nerve stimulation (tVNS) and myofascial release exercises in patient wiht chronic subjective tinnitus. Participants will be randomly assigned into three groups: (1) tVNS group, (2) Myofascial exercise group, and (3) Control group receiving standart medical care. The primary outcome is change in tinnitus severity measured by the Tinnitus Handicap Inventory (THI). Secondary outcomes include tinnitus loudness Visual Analouge Scale for Tinnitus (VAS), sleep quality Pitsburgh Sleep Quality Index (PSQI) and audiometric findings.

DETAILED DESCRIPTION:
Tinnitus is a common and distressing condition that significantly impairs quality of life. Recent studies suggest that neuromdulation techniques such as vagus nerve stimulation and physical interventions targeting myofascial structures may reduce tinnitus severity. However, evidence remains limited, and comparative effectiveness of these approaches is not well established.

This single-center randomized controlled trial will compare the effects of transcutaneous vagus nerve stimulation (tVNS) and myofascial release exercises with a control group receiving only medical treatment. A total of 45 participants with chronic subjective tinnitus will be recruited. Participants will be randomized into three groups and receive 10 intervention sessions over three weeks.

The tVNS group will receive transcutaneous stimulation of the auricular branch of the vagus nerve using a TENS (Everyway N604, Taiwan) device. The myofascial group will undergo guided myofascial release targeting cervical muscles in addition to medical treatment. The control group will continue their medical treatment without additional interventions.

The primary outcome measure will be change in tinnitus-related handicap using the Tinnitus Handicap Inventory (THI). Secondary outcomes will include tinnitus loudness assesed by a Visual Analogue Scale for Tinnitus (VAS), sleep quality measured by the Pittsburgh Sleep Quality Index (PSQI) and audiometric assesments.

The findings from this trial may provide new insights into non-farmacological rehabiliation strategies for tinnitus and clarify the role of neuromodulation compared with physical therapy inreventions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic subjective tinnitus (>6 months)
* Ability to understand and provide written informed consent
* Willingness to comply with study procedures and intervention schedule
* Resistant for medical treatment for subjective tinnitus
* Impacted daily living by tinnitus

Exclusion Criteria:

* Diagnoses such as auditory hallucinations, Meniere's disease, vestibular tumor, vertigo, or sudden hearing loss
* Trauma or surgical interventions involving the neck, jaw, or head within the 6 months
* Epilepsy or presence of a cardiac pacemaker (contraindication for tVNS)
* History of acute psychiatric disorders
* Use of ototoxic medications
* Physical limitations that prevent participation in exercise interventions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Change in tinnitus severity | Baseline to post-intervention (3 weeks)
  Measured using the Tinnitus Handicap Inventory (THI), which assesses the impact of tinnitus on daily functioning.

SECONDARY OUTCOMES:
Tinnitus Loudness | Baseline to post-intervention (3 weeks)
  Assessed using Visual Analogue Scale for Tinnitus (VAS)
Sleep quality | Baseline to post-intervention (3 weeks)
  Measured using the Pittsburgh Sleep Quality Index (PSQI).
Audiometric measures | Baseline to post-intervention (3 weeks)
  Pure-tone audiometry to assess hearing tresholds across frequencies

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan ALTUNTAŞ YILMAZ, PhD, Principal Investigator — Necmettin Erbakan University Nezahat Kelesoglu Faculty of Health Sciences; Mehmet Akif DUNDAR, PhD, Study Director — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University Meram Faculty of Medicine, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Demographics, efficacy outcomes, safety data
Supporting Information: Study Protocol, SAP
Time Frame: 12 months after study completion-5 years after completion
Access Criteria: Data available upon request to qualified researchers for scientific purposes. Requests should be sent to the Principal Investigator via the contact page below. Data will be shared after signing a data use agreement.
URL: https://www.erbakan.edu.tr/tr/akademik-personel/5196-NESL%C4%B0HAN-ALTUNTA%C5%9E%20YILMAZ

REFERENCES:
- [Background] Rocha CB, Sanchez TG. Efficacy of myofascial trigger point deactivation for tinnitus control. Braz J Otorhinolaryngol. 2012 Dec;78(6):21-6. doi: 10.5935/1808-8694.20120028. PMID 23306563
- [Background] Yakunina N, Nam EC. Direct and Transcutaneous Vagus Nerve Stimulation for Treatment of Tinnitus: A Scoping Review. Front Neurosci. 2021 May 28;15:680590. doi: 10.3389/fnins.2021.680590. eCollection 2021. PMID 34122002
- See also: This webpage provides information about Dr. Neslihan Altuntaş Yılmaz, a faculty member at the Department of Physiotherapy and Rehabilitation, Necmettin Erbakan University. Researchers interested in accessing individual participant data (IPD) from this cl — https://www.erbakan.edu.tr/tr/akademik-personel/5196-NESL%C4%B0HAN-ALTUNTA%C5%9E%20YILMAZ